CLINICAL TRIAL: NCT02765009
Title: Effects of Fluid Balance Control in Critically Ill Patients: A Multicenter Randomized Study
Brief Title: Effects of Fluid Balance Control in Critically Ill Patients
Acronym: POINCARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2015-A00662-47
Record Dates: First submitted 2016-04-29; First posted 2016-05-06 (Estimated); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Fluid Shifts; Critical Care
Keywords: Fluid overload; Multiple organ failure; Diuretics; Fluid restriction; Body weight
MeSH Terms: conditions — Edema; Multiple Organ Failure; Body Weight | interventions — Diuretics; Hydrochlorothiazide; Bumetanide; Furosemide; Albumins; Ultrafiltration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Usual care provided according to the ward policy. Patients have to be weighed at least on admission (day 0), day 7 and day 14.
- Strategy (Experimental): Patients have to be weighed every day. Use of an algorithm based on weight changes from day 2 to day 14 in order to reduce weight gain (fluid overload) using diuretics, fluid restriction,albumin, and ultrafiltration (the latter when ongoing renal replacement)
  Interventions: Drug: diuretics; Drug: albumin; Other: fluid restriction; Device: renal replacement

INTERVENTIONS:
Drug: diuretics — Used to reduce fluid overload as evidenced by weight gain
  Other Names: hydrochlorothiazide; bumetanide; furosemide
  Arms: Strategy
Drug: albumin — Used to reduce fluid overload in addition with diuretics in hypoalbuminemic patients
  Arms: Strategy
Other: fluid restriction — Used to reduce fluid overload
  Arms: Strategy
Device: renal replacement — Used to reduce fluid overload in patients with renal replacement
  Other Names: ultrafiltration
  Arms: Strategy

SUMMARY:
Most ICU patients develop a positive fluid balance, mainly during the two first weeks of their stay. The causes are multifactorial: a reduced urine output subsequent to shock state, positive pressure mechanical ventilation, acute renal failure, post-operative period of major surgical procedures, and simultaneous fluid loading to maintain volemia and acceptable arterial pressure. Additionally, the efficacy of fluid loading is frequently suboptimal, in relation to severe hypoalbuminemia and inflammatory capillary leakage. This results usually in a cumulated positive fluid balance of more than 10 litres at the end of the first week of stay. A high number of studies have showed that such a positive fluid balance was an independent factor of worse prognosis in selected populations of ICU patients: acute renal failure, acute respiratory distress syndrome (ARDS), sepsis, post-operative of high risk surgery. However, little is known about the putative causal role of positive fluid balance by itself on outcome. However, in two randomized controlled studies in patients with ARDS, a strategy of fluid balance control has been demonstrated to reduce time under mechanical ventilation and ICU length of stay with no noticeable adverse effects. Although avoiding fluid overload is now recommended in ARDS management, there is no evidence that this approach would be beneficial in a more general population of ICU patients (i.e. with sepsis, acute renal failure, mechanical ventilation). In addition, fluid restriction -mainly if applied early could be deleterious in reducing both tissue oxygen delivery and perfusion pressure. There is a place for a prospective study comparing a "conventional" attitude based on liberal fluid management throughout the ICU stay with a restrictive approach aiming at controlling fluid balance, at least as soon as the patient circulatory status is stabilized. The latter approach would use a simple algorithm using fluid restriction and diuretics based on daily weighing, a common procedure in the ICU, probably more reliable than cumulative measurement of fluid movements in patients whose limits have been underlined.

ELIGIBILITY:
Inclusion Criteria:

* Patients under mechanical ventilation, admitted for > 48h and <72h and no discharge planned for the next 24h

Exclusion Criteria:

* Age < 18 years
* Failure to weigh the patient
* Multiple trauma
* Transfer from another ICU with a previous stay > 24h
* High probability of withdrawing treatment for ethical purposes within 7 days
* Pregnancy
* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1411 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2020-05-25 (Actual)

PRIMARY OUTCOMES:
All-cause mortality at 60 days after inclusion | 60 days
  Vital status collected 60 days after admission; if the patient was dead at the time of assessment, date of death was collected

SECONDARY OUTCOMES:
Fluid balance control at day 7 | 7 days
  Mean differences of patient body weight between Day 7 and admission (Day 0)
Fluid balance control at day 14 | 14 days
  Mean differences of patient body weight between Day 14 and admission (Day 0)
All-cause mortality at 28-day after inclusion | 28 days
  Vital status collected 28 days after admission
All-cause in-hospital mortality | Up to 24 weeks
  Death during the hospital stay where the patient was included in the study
All-cause mortality at 365 days after inclusion | 365 days
  Vital status collected one year after admission
Survival time period at Day 60 | 60 days
  Time-related mortality, calculated from admission to the date of death
Survival time period at Day 365 | 365 days
  Time-related mortality, calculated from admission to the date of death
Global end-organ damage assessment | 28 days
  Time-related changes of Sequential Organ Failure Assessment (SOFA score): SOFA is a score of organ failure with 6 subscales on organ dysfunction: respiratory, neurological, cardiovascular,hepatic,renal and coagulation. Each ranges from 0 to 4 and the total SOFA score is the sum of each subscale ; increasing severity from 0 (normal) to 24(moribund). Values of SOFA score are tightly correlated with mortality.
Dependence on vasopressor drugs | 28 days
  Cumulated number of vasopressor-free days alive from day 0 to day 28
Dependence on mechanical ventilation | 28 days
  Cumulated number of ventilator-free days alive from day 0 to day 28
Dependence on renal replacement therapy | 60 days
  Cumulated number of renal replacement-free days alive from day 0 to day 60
Cumulated number of pre-defined adverse events | 14 days
  Pre-defined adverse events include Systolic arterial pressure< 90 mm Hg, kalemia < 2,8 ,mmol/L, natremia >155 mmol/L, "injury" level of renal dysfunction (RIFLE scale), acute ischemic events (myocardial infarction, mesenteric ischemia)

CONTACTS AND LOCATIONS:
Overall Officials: El Mehdi Siaghy, Study Director — Central Hospital, Nancy, France
Locations (11):
- France (11):
  - Hopital Nord Franche-Comté, Belfort
  - Centre Hospitalier Universitaire, Dijon
  - Centre Hospitalier Universitaire, Lyon
  - Centre Hospitalier Régional, Metz
  - Centre Hospitalier Régional et Universitaire, Nancy
  - Groupe Hospitalier Saint Joseph, Paris
  - Centre Hospitalier intercommunal, Poissy
  - Centre Hospitalier Régional et Universitaire, Strasbourg
  - CentreHospitalier Régional et universitaire, Strasbourg
  - Centre Hospitalier Régional, Thionville
  - Centre Hospitalier, Verdun

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agrinier N, Monnier A, Argaud L, Bemer M, Virion JM, Alleyrat C, Charpentier C, Ziegler L, Louis G, Bruel C, Jamme M, Quenot JP, Badie J, Schneider F, Bollaert PE. Effect of fluid balance control in critically ill patients: Design of the stepped wedge trial POINCARE-2. Contemp Clin Trials. 2019 Aug;83:109-116. doi: 10.1016/j.cct.2019.06.020. Epub 2019 Jun 29. PMID 31260794
- [Derived] Buzzi M, Ricci L, Gibot S, Argaud L, Badie J, Bruel C, Charpentier C, Outin H, Louis G, Monnier A, Quenot JP, Schneider F, Minary L, Agrinier N. Implementation of a fluid balance control strategy in critically ill patients: POINCARE-2 trial process evaluation. BMC Med Res Methodol. 2024 Jul 24;24(1):160. doi: 10.1186/s12874-024-02288-1. PMID 39048932
- [Derived] Mansouri A, Buzzi M, Gibot S, Charpentier C, Schneider F, Louis G, Outin H, Monnier A, Quenot JP, Badie J, Argaud L, Bruel C, Soudant M, Agrinier N; the POINCARE-2 group. Fluid balance control in critically ill patients: results from as-treated analyses of POINCARE-2 randomized trial. Crit Care. 2023 Nov 6;27(1):426. doi: 10.1186/s13054-023-04701-5. PMID 37932787
- [Derived] Bollaert PE, Monnier A, Schneider F, Argaud L, Badie J, Charpentier C, Meziani F, Bemer M, Quenot JP, Buzzi M, Outin H, Bruel C, Ziegler L, Gibot S, Virion JM, Alleyrat C, Louis G, Agrinier N. Fluid balance control in critically ill patients: results from POINCARE-2 stepped wedge cluster-randomized trial. Crit Care. 2023 Feb 21;27(1):66. doi: 10.1186/s13054-023-04357-1. PMID 36810101